CLINICAL TRIAL: NCT05535751
Title: Cefepime vs. Carbapenems for Treating AmpC β-lactamase-producing Enterobacteriaceae Bloodstream Infections
Acronym: CARBAPENEM
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8660
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Bacteremia
Keywords: Bacteremia; Cefepime; carbapenems; AmpC β-lactamase; enterobacteriaceae bloodstream infections
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recent international recommendations suggest the use of carbapenem rather than cefepime in this situation, but with a low level of evidence, given the few existing studies. As cefepime is a less broad-spectrum antibiotic than carbapenems, its use would limit the selection of multidrug-resistant bacteria.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years of age)
* managed within a study center for high-grade cephalosporinase-producing bacteremia
* Not objecting to the reuse of their health data for scientific research purposes.

Exclusion Criteria:

* Patient who has expressed opposition to the reuse of their data for scientific research purposes.
* Resistance to Cefepime or carbapenems
* Multiple bacteremia
* Treatment with a molecule other than Cefepime or carbapenem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years of age) managed within a study center for high-grade cephalosporinase-producing bacteremia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | 30 days after infection

CONTACTS AND LOCATIONS:
Locations (1):
- Service des maladies infectieuses et tropicales - CHU de Strasbourg - France, Strasbourg, France